CLINICAL TRIAL: NCT02650219
Title: Prevalence of Autoantibodies in the Gaucher Disease and the Role of CD1 Molecules in Immune Manifestations of This Disease
Brief Title: Auto-antibodies Prevalence and CD1 Role in Gaucher Disease
Status: Completed | Type: Observational
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Christine Serratrice, MD head of internal medicine department, Hospital St. Joseph, Marseille, France
Other Study IDs: ID-RCB 2010-A00315-3
Record Dates: First submitted 2016-01-05; First posted 2016-01-08 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-02

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Genetic Linkage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- gaucher disease type 1: Inclusion criteria:
  * Adult patients >= 18 years old
  * Gaucher disease type 1, proved by low betaglucosidase, with or without treatment
  * Patients must have read, understood and signed informed consent. intervention : genetic analyses
  Interventions: Genetic: genetic analyses
- Control: healthy subjects intervention: genetic analyses
  Interventions: Genetic: genetic analyses

INTERVENTIONS:
Genetic: genetic analyses

SUMMARY:
Hypergammaglobulinaemia is frequently observed in type 1 Gaucher disease (GD1), being either polyclonal or monoclonal gammopathies. Polyclonal hypergammaglobulinemia may be related to the presence of autoantibodies. The clinical significance of such antibodies is questioned in Gaucher disease (GD), as some cases of immunologic thrombocytopenia and autoimmune hemolytic anemia have also been reported.

Objectives:

To evaluate the prevalence of autoantibodies and autoimmune diseases in GD1 patients, we conducted a multicenter national study. The investigators investigated whether there was a link between splenectomy, genotype, therapeutic options and the presence of these autoantibodies.They also investigated whether there was a correlation with some clinical manifestations of GD1

ELIGIBILITY:
for GD1 patients

Inclusion Criteria:

* Adult patients >= 18 years old
* Gaucher disease type 1, proved by low betaglucosidase, with or without treatment
* Patients must have read, understood and signed informed consent.

Exclusion Criteria:

* Under 18 years old
* Pregnant or breast-feeding
* Patients under administrative control
* Prisoners
* Patients without social rights
* Emergency hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 40 GD1 patients and 20 healthy volunteers (control group) were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Serratrice, MD, Principal Investigator — St joseph France
Locations (11):
- France (11):
  - Internal Medicine Department, Hôpital Minjoz,, Besançon
  - Intensive Care Department, Hôpital Pellegrin,, Bordeaux
  - Internal Medicine Department, Hôpital Beaujon,, Clichy
  - Internal Medicine and Clinical Immunology Department, CHU,, Dijon
  - Internal Medicine Department, Catholic University,, Lille
  - Internal Medicine Department, CHU, Nantes, Nantes
  - Internal Medicine and Rheumatology Department, Hôpital La Croix Saint Simon,, Paris
  - Internal Medicine Department, CHU la Pitié Salpêtrière,, Paris
  - 13 Internal Medicine Department, CHU,, Rouen
  - CHRU de Tours, Université François Rabelais, INSERM 1069,, Tours
  - Internal Medicine and Immunology Department, CHU Hôpital Brabois,, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: from January 2010 to April 2011, 40 GD1 patients and 20 healthy volunteers (control group) were included in the study in the 12 inclusions centers (medical clinic or hopsital)
Groups:
- Gaucher Disease Type 1: Inclusion criteria:
  * Adult patients >= 18 years old
  * Gaucher disease type 1, proved by low betaglucosidase, with or without treatment
  * Patients must have read, understood and signed informed consent. intervention : genetic analyses
  genetic analyses
- Control: healthy subjects intervention: genetic analyses
  genetic analyses
Period: Overall Study
Arm/Group | Gaucher Disease Type 1 | Control
Started | 40 | 20
Completed | 40 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gaucher Disease Type 1 | Control | Total
Number analyzed (Participants) | 40 | 20 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 17 | 48
  >=65 years | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 52.4 (13.4) | 47.3 (15.4) | 50.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 18 | 7 | 25
Region of Enrollment [Number; unit: participants]
  France | 40 | 20 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With GD Diagnosis Confirmed by : Enzyme Testing of acidβ-glucosidase Activity Activity <15% in Blood Leucocytes Completed When Necsssary by GB1 Mutation Analyses (Analyses From Samples)
Description: acidβ-glucosidase enzyme testing : a lower than 15% of mean normal activity is considered to be diagnostic.
  Decreased enzyme levels will often be confirmed by genetic testing. Numerous different mutations occur; GB1 mutation analyses is sometimes necessary to confirm the diagnosis.
Time Frame: baseline
Measure: Number; unit: participant
Arm/Group | Gaucher Disease Type 1 | Control
Number analyzed (Participants) | 40 | 20
participant | 40 | 0

2. Secondary Outcome: Number of Patients With : Splenectomy and/or Bone Events and/or Pulmonary Hypertension and/or Specific Treatment and Non-specific (Medical History,Physiological Parameters and Questionnaire)
Description: data available from medical record of the patients
Time Frame: Baseline
Population: splenectomy testing
Measure: Number; unit: participants
Arm/Group | Gaucher Disease Type 1 | Control
Number analyzed (Participants) | 40 | 20
participants | 15 | 0

3. Secondary Outcome: Number of Patients With : Photosensitivity and/or Raynaud Phenomenon and/or Sicca Syndrome and/or Arthralgia and/or Arthritis and/or Thrombosis (Medical History and Questionnaire)
Description: Features usually associated with auto immune disease- data available from medical record of the patients
Time Frame: Baseline
Reporting Status: Not Posted

4. Secondary Outcome: Number of Patients With : Antinuclear and/or Anti-SSa and/or Anti-SSb and/or Anti-RNP and/or Anti-DNA and/or Anti-Sm and/or Anticardiolipid and/or Anti β2Gp1 and/or Antiganglioside Autoantibodies (Genetics Analyses From Blood Samples)
Description: data available from biological analyses (blood samples)
Time Frame: baseline
Population: antinuclear autoantibodies
Measure: Number; unit: participants
Arm/Group | Gaucher Disease Type 1 | Control
Number analyzed (Participants) | 40 | 20
participants | 10 | 3

ADVERSE EVENTS:
Arm/Group | Gaucher Disease Type 1 | Control
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/20
Other Adverse Events (participants affected / at risk) | 0/40 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No